CLINICAL TRIAL: NCT05779722
Title: The Effect of a Vapor Barrier in Combination With Active External Rewarming for Patients
Brief Title: The Effect of a Vapor Barrier in Combination With Active External Rewarming for Patients With Accidental Hypothermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 566433
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Hypothermia, Accidental
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: The study will use a crossover design on where research participants will undergo repetitions of the same scenario with different interventions in order to serve as their own control.
  We intend to perform the experiments in an outdoor laboratory in order to achieve the most realistic conditions possible. The experiments will be conducted in Hemsedal, Norway in our "Mountain Lab", a climate chamber built inside a snow cave.
  Before the start of the experiment, the research participants will be positioned in a supine position in the snow cave on an insulated stretcher in wet clothes saturated with a standardized amount of water. They will stay in this position for 45 minutes to allow for a drop in the skin temperature without a drop in core body temperature. After 45 minutes, the research participant will be randomised into one of two scenarios, intervention or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): wrapping the participants in a vapor barrier as the inner layer (intervention),
  Interventions: Device: Vapor barrier
- No intervention (No Intervention): without the vapor barrier to serve as a negative control

INTERVENTIONS:
Device: Vapor barrier — Vapor barrier
  Arms: Intervention

SUMMARY:
Most guidelines recommend the use of a vapor barrier when wrapping and isolating hypothermic patients from the environment, and this is especially important if the patient is wearing wet clothing. The vapor barrier will contain moisture evaporated from the wet clothes of the patient and increase the humidity. Once the humidity levels reach 100%, the evaporation and thereby the evaporative heat loss will stop. The theory is that the addition of a vapor barrier will reduce the amount of heat loss and contribute to more efficient rewarming of wet, hypothermic patients. We aim to investigate how much more efficient a wrapping model with active external rewarming is with the addition of a vapor barrier.

DETAILED DESCRIPTION:
The study will use a crossover design on where research participants will undergo repetitions of the same scenario with different interventions in order to serve as their own control. The research participants will be healthy volunteers providing both oral and written consent.

We intend to perform the experiments in an outdoor laboratory in order to achieve the most realistic conditions possible. The experiments will be conducted in Hemsedal, Norway in our "Mountain Lab", a climate chamber built inside a snow cave.

Before the start of the experiment, the research participants will be positioned in a supine position in the snow cave on an insulated stretcher in wet clothes saturated with a standardized amount of water.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* any cronic sickness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-03-17 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Skin temperature | 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn Nedrebø, PhD, Study Director — Research director
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mydske S, Brattebo G, Osteras O, Wiggen O, Assmus J, Thomassen O. Effect of a vapor barrier in combination with active external rewarming for cold-stressed patients in a prehospital setting: a randomized, crossover field study. Scand J Trauma Resusc Emerg Med. 2024 Apr 25;32(1):35. doi: 10.1186/s13049-024-01204-2. PMID 38664809